CLINICAL TRIAL: NCT06060197
Title: Caregiver-reported Economic Burden and Quality of Life Impact of Monocarboxylate Transporter 8 (MCT8) Deficiency
Brief Title: MCT8 Deficiency Caregiver Study
Status: Completed | Type: Observational
Sponsor: Rare Thyroid Therapeutics International AB (Industry)
Collaborators: Vitaccess Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 4253-09-2021
Record Dates: First submitted 2023-08-11; First posted 2023-09-29 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Monocarboxylate Transporter 8 (MCT8) Deficiency; Allan-Herndon-Dudley Syndrome
Keywords: MCT8 deficiency; caregiver; economic burden; HRQoL; EQ-5D-5L; PROs
MeSH Terms: conditions — Allan-Herndon-Dudley syndrome; Financial Stress

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Caregivers face many responsibilities outside of their role as a friend or parent, which can lead to emotional, financial, social, and professional challenges. To better understand the impact of MCT8 deficiency on caregivers, Egetis Therapeutics are conducting an online survey for adult caregivers of persons living with the MCT8 deficiency.

DETAILED DESCRIPTION:
Understanding the impact of MCT8 deficiency on caregivers and patients is key to facilitating evidence-based policy interventions and identifying better treatments and treatment practices that take full account of the actual environment in which care is delivered.

This study will address the gap in research about the wider impact of MCT8 deficiency by exploring the caregiver-reported economic burden and health-related quality of life (HRQoL) impact of the disease. Adult caregivers will report HRQoL outcomes for themselves and the person with MCT8 deficiency that they care for, as affected patients have limited cognitive function and communication abilities and cannot report the information themselves.

The results from this study will provide insight into the economic and HRQoL impact of MCT8 deficiency, as reported by caregivers, in the UK, US, Canada, France, Netherlands, Spain, Australia, Italy, and Germany.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Resident in the UK, US, Canada (except Newfoundland & Labrador and Alberta), France, Netherlands, Spain, Australia, Italy, and Germany
* Main caregiver to a person diagnosed with MCT8 deficiency

Exclusion Criteria:

* Paid caregivers to a person diagnosed with MCT8 deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who are the main caregiver to a person diagnosed with MCT8 deficiency or Allan-Herndon-Dudley syndrome and regularly provide a significant amount of help to them.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Quantify the economic burden of caring for a patient with MCT8 deficiency using bespoke questions | once, at enrolment
  Economic burden will be assessed by using bespoke questions on the time spent providing care and impact on caregiver's family and work circumstances.
Quantify the cost of caring for a patient with MCT8 deficiency using bespoke questions | once, at enrolment
  Costs will be assessed by using bespoke questions on the caregiver's employment income, costs of travel/transport, contributions to the costs of treatments and other costs of care.
Quantify the health-related quality of life (HRQoL) burden of caring for a patient with MCT8 deficiency using the EQ-5D-5L | once, at enrolment
  The impact on the caregiver's wellbeing will be assessed using the EQ-5D-5L, which comprises two parts. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with 5 levels (1 - no problems, 2 - slight problems, 3 - moderate problems, 4 - severe problems, and 5 - extreme problems). The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state.
  The EQ Visual Analogue Scale (EQ-VAS) records the respondent's self-rated health on a vertical scale with endpoints labelled 100, representing 'the best health you can imagine' and 0, 'the worst health you can imagine'. Higher scores represent better self-perceived health.
Quantify the health-related quality of life (HRQoL) burden of caring for a patient with MCT8 deficiency using the PedsQL | once, at enrolment
  The impact on the caregiver's family will be assessed using the Pedriatric Quality of Life Inventory (PedsQL™) Family Impact Module. The PedsQL™ has 36 items broken down into 7 subdomains of physical, emotional, social, and cognitive functioning, communication, and worry as well as family daily activities and family relationships. A 5-point response scale is utilized (0 = never a problem; 4 = always a problem). Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), so that higher scores indicate better functioning (less negative impact).

SECONDARY OUTCOMES:
Describe the social and demographic characteristics of patients and caregivers | once, at enrolment
  This will be assessed using the caregiver age, sex, relationship to the person with MCT8 deficiency, household information and caring responsibilities. Limited data will also be analyzed on the profile of the person being cared for with MCT8 deficiency, specifically patient's age, functioning (physical and communication), tests done related to MCT8 deficiency, the range of medical professionals seen for treatment, and frequency and length of hospital stays.
Investigate the experiences of caregivers providing care and support to patients affected by MCT8 deficiency | once, at enrolment
  Caregiver experience will be assessed using responses provided to bespoke questions on family circumstances, other caring responsibilities, impact of caregiving on their sleep, domestic and professional support at home. All bespoke questions are categorical variables with various response options.
Provide additional evidence on the HRQoL of patients with MCT8 deficiency across health states using the EQ-5D-5L proxy version 1 | once, at enrolment
  EQ-5D-5L proxy version 1 will be captured from the caregiver (the proxy) to rate the person with MCT8 deficiency's health-related quality of life in their (the proxy's) opinion. The instrument comprises two parts. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with 5 levels (1 - no problems, 2 - slight problems, 3 - moderate problems, 4 - severe problems, and 5 - extreme problems). The digits for 5 dimensions can be combined in a 5-digit number describing the health state of the person the respondent is reporting on.
  The EQ Visual Analogue Scale (EQ-VAS) records how the respondent would rank the person's health on a vertical scale with endpoints labelled 100, representing 'the best health you can imagine' and 0, 'the worst health you can imagine'. Higher scores represent better self-perceived health.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Larkin, PhD, Principal Investigator — Vitaccess Limited
Locations (1):
- Vitaccess Ltd, Oxford, Oxfordshire, United Kingdom